CLINICAL TRIAL: NCT03841656
Title: Influence of Periodontal Care Response on Implant Treatment Outcomes at Long-term
Brief Title: Influence of Gum Disease Treatment on Long-term Dental Implant Success
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 67RC001
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PARORISKIMPLANT — Patients attending periodontal and implant treatment at the Department of Periodontology of the Dental Faculty at Strasbourg, France, between 2000-2015.

SUMMARY:
The aim of this study is to evaluate the influence of periodontal care response on long term dental implant success. Investigator's hypothesis is that patients who do not well respond to periodontal care have more chance to develop peri-implant complications at long-term. The second purpose of this study is to evaluate the influence of other local, systemic, behavioral, and implant's related risk factors

ELIGIBILITY:
Inclusion Criteria:

Patient attending supporting periodontal therapy with at least one implant placed for more than 3 years

* Patient with more than 12 teeth at baseline
* Patient with demographic, periodontal, implant data recording
* patient aged >30 years at Baseline

Exclusion criteria:

* Patient needed antibiotic prophylaxis
* Uncontrolled diabetes
* Systemic inflammatory or autoimmune diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient attending periodontal and implant treatment at the Department of Periodontology of the Dental Faculty at Strasbourg, France, between 2000-2015.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Presence of peri-implantitis as measured by probing depth | At least 3 years after dental implant placement
  The implant has a probing depth more than or equal to 4 mm
Presence of peri-implantitis as measured by erythema | At least 3 years after dental implant placement
  The implant has bleeding on probing
Presence of peri-implantitis as measured by radiographic bone loss | At least 3 years after dental implant placement
  The implant has a radiographic bone loss when compared to previous radiographs

SECONDARY OUTCOMES:
Implant survival | At least 3 years after dental implant placement
  presence of implant on arch Peri-implant mucositis: presence of bleeding on probing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papalou I, Vagia P, Cakir A, Tenenbaum H, Huck O, Davideau JL. Influence of Periodontitis, Implant, and Prosthesis Characteristics on the Peri-Implant Status: A Cross-Sectional Study. Int J Dent. 2022 Feb 7;2022:9984871. doi: 10.1155/2022/9984871. eCollection 2022. PMID 35178092